CLINICAL TRIAL: NCT03668548
Title: The Effects of 10-week Leucine Supplementation on Muscle Growth, Body Composition, Metabolism, Inflammation and Wellbeing of Adolescents and Young Adults With Cerebral Palsy
Brief Title: 10-week Leucine Supplementation in Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: St Mary's University College (Other)
Collaborators: University of Gloucestershire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC.18.85.7
Record Dates: First submitted 2018-08-20; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Cerebral Palsy; Cerebral Palsy, Mixed; Cerebral Palsy Ataxic
MeSH Terms: conditions — Cerebral Palsy; Cerebral Palsy, Ataxic, Autosomal Recessive | interventions — Leucine; Amino Acids

STUDY DESIGN:
Intervention Model Description: The study will be a randomised controlled pilot trial. Participants will complete testing at baseline and after 10 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties will be masked from the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leucine group (Experimental): To receive leucine on a daily basis for 10 weeks
  Interventions: Dietary Supplement: Leucine
- Control group (Placebo Comparator): To receive a placebo supplement on a daily basis for 10 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Leucine — 192 mg/kg body mass/day
  Other Names: Amino Acid
  Arms: Leucine group
Dietary Supplement: Placebo — A taste and calorie-matched placebo
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the effects of 10-weeks leucine supplementation on muscle growth, metabolism, body composition, inflammation and wellbeing in adolescents and young adults with CP.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is caused by damage to the developing brain and descending pathways, leading to altered patterns of growth and development. Those with CP may encounter early symptoms of paresis and spasticity, leading to progressive secondary musculoskeletal complications, including increased muscle atrophy and abnormal growth of contractile and non-contractile tissue. This causes significant weakness of the muscle and compromises daily motor function, leading to substantial declines in activities of daily living and independence. As such, interventions aimed at increasing muscle mass or preventing muscle atrophy for those with CP must be established. It is well established that dietary protein ingestion stimulates protein synthesis and inhibits proteolytic pathways, resulting in a positive protein balance and net muscle mass gain. In particular, leucine (a branched chain amino acid; BCAA), has been used to facilitate protein synthesis and muscle growth. Leucine also has anti-inflammatory roles, some of which are central in origin and have been shown to effect mood and features of wellbeing. However, there has been no investigation of the effects of leucine supplementation on any of these parameters in CP. Therefore, the purpose of this study is to assess the effects of 10-weeks leucine supplementation on muscle growth, metabolism, body composition, inflammation and wellbeing in adolescents and young adults with CP.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of spastic cerebral palsy
* Aged 12-22 years

Exclusion Criteria:

* Orthopaedic surgery of the upper-limbs in the past 12 months
* Botulinum toxin type A injections in the past 6 months
* Serial casting in the past 6 months
* Insufficient cognitive understanding to comply with the assessment procedures and intervention
* Liver and/or kidney dysfunction

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-10-22 (Estimated); Study Completion 2018-10-22 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle volume | 10 weeks
  Change in biceps brachii volume

SECONDARY OUTCOMES:
Resting metabolic rate | 10 weeks
  Change in resting energy expenditure and substrate metabolism
Perceptual well-being questionnaire | 10 weeks
  Change in a composite measure of five different wellbeing sub-components
Systemic inflammation (C-Reactive protein; C-RP) | 10 weeks
  Change in C-RP
Skeletal muscle strength | 10 weeks
  Change in the biceps brachii force production

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Theis, PhD, Principal Investigator — University of Gloucestershire
Locations (2):
- United Kingdom (2):
  - University of Gloucestershire, Cheltenham, Gloucestershire
  - St Marys Umiversity College, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Theis N, Brown MA, Wood P, Waldron M. Leucine Supplementation Increases Muscle Strength and Volume, Reduces Inflammation, and Affects Wellbeing in Adults and Adolescents with Cerebral Palsy. J Nutr. 2021 Jan 4;151(1):59-64. doi: 10.1093/jn/nxaa006. PMID 31965179